CLINICAL TRIAL: NCT01930045
Title: A Study to Evaluate the Effect of Staggered Dosing of a Magnesium/Aluminum Antacid on Raltegravir Pharmacokinetics in HIV-Infected Subjects on a Raltegravir-Containing Regimen
Brief Title: A Pharmacokinetic Study to Evaluate the Effect of MAALOX on Raltegravir (MK-0518) in Human Immunodeficiency Virus (HIV)-Infected Participants (MK-0518-295)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0518-295
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; aluminum hydroxide, magnesium hydroxide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ralt→MAL4Ralt→Ralt4MAL→MAL6Ralt→Ralt6MAL (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: Raltegravir (Ralt) alone in Period 1, MAALOX (MAL) followed 4 hrs later by Ralt in Period 2, Ralt followed 4 hrs later by MAL in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)
- MAL4Ralt→Ralt4MAL→Ralt→MAL6Ralt→Ralt6MAL (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: MAL followed 4 hrs later by Ralt in Period 1, Ralt followed 4 hrs later by MAL in Period 2, Ralt alone in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)
- Ralt4MAL→Ralt→MAL4Ralt→MAL6Ralt→Ralt6MAL (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: Ralt followed 4 hrs later by MAL in Period 1, Ralt alone in Period 2, MAL followed 4 hrs later by Ralt in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)
- Ralt→Ralt4MAL→MAL4Ralt→Ralt6MAL→MAL6Ralt (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: Ralt alone in Period 1, Ralt followed 4 hrs later by MAL in Period 2, MAL followed 4 hrs later by Ralt in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)
- MAL4Ralt→Ralt→Ralt4MAL→Ralt6MAL→MAL6Ralt (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: MAL followed 4 hrs later by Ralt in Period 1, Ralt alone in Period 2, Ralt followed 4 hrs later by MAL in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)
- Ralt4MAL→MAL4Ralt→Ralt→Ralt6MAL→MAL6Ralt (Experimental): Part 1 was comprised of periods 1, 2 and 3; Part 2 was comprised of periods 4 and 5; with each study period separated by a washout period of at least 2 days. Part 1 was separated from Part 2 by a Pause. Each period had single oral dose treatments as follows: Ralt followed 4 hrs later by MAL in Period 1, MAL followed 4 hrs later by Ralt in Period 2, Ralt alone in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
  Interventions: Drug: Raltegravir (ISENTRESS™); Drug: MAALOX (MAL)

INTERVENTIONS:
Drug: Raltegravir (ISENTRESS™) — Raltegravir 400 mg oral tablet once every 12 hours. Participants will continue with their other prescribed antiretroviral agents throughout the study.
Drug: MAALOX (MAL) — MAL (or generic equivalent) 20 mL oral single dose on Day 1
  Other Names: MAALOX® MS

SUMMARY:
This study evaluated the effect of single doses of a magnesium/aluminum antacid (MAALOX) given 4 and 6 hours before or after administration of raltegravir, on the pharmacokinetics of raltegravir in human immunodeficiency virus (HIV)-infected participants. The study consisted of Part 1 (Periods 1, 2, and 3) and Part 2 (Periods 4 and 5), with each study period separated by a washout period of at least 2 days; Part 1 was separated from Part 2 by a Pause. Each study period had a duration of ≥2 days, and paused for evaluation of Part 1 pharmacokinetics results before continuing to Part 2. The same participants participated in Parts 1 and 2. The primary hypothesis tested (in Part 1) was that raltegravir plasma concentration 12 hours after administration (C 12 hrs) would not differ significantly from raltegravir C 12 hrs when antacid is administered 4 hours before or 4 hours after raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* On a stable raltegravir dose as part of a stable antiretroviral regimen for ≥1 month before the study
* If female, is not pregnant or breast feeding
* Body mass index ≤32 kg/m^2

Exclusion Criteria:

* Mentally or physically incapacitated, has significant emotional problems, or history of clinically significant psychiatric disorder within ≤10 years
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or disease (excluding HIV)
* History of gastric bypass surgery
* History of cancer, except adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated ≥10 years before the study
* History of chronic diarrhea within ≤3 months before the study
* History of significant multiple and/or severe allergies (food, drug, latex), or had an anaphylactic reaction or significant intolerability to drugs or food
* Had major surgery or donated or lost ≥1 unit of blood (500 mL) ≤4 weeks before the study
* Participated in another investigational trial ≤4 weeks before the study
* Taking rifampin or is unable to refrain from the use of 1) any proton pump inhibitor from 2 weeks before and throughout the study, or 2) any histamine H2-blockers, antacids, calcium supplements, or multivitamins from 2 weeks before and throughout the study
* Consumes >3 glasses of alcoholic beverages per day
* Consumes excessive amounts of caffeine beverages (coffee, tea, cola, energy drinks, or other caffeinated drinks) per day
* Currently uses or has a history of drug abuse within ≤6 months before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2013-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0518-295&kw=0518-295&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: Raltegravir (Ralt) alone in Period 1, MAALOX (MAL) followed 4 hrs later by Ralt in Period 2, Ralt followed 4 hrs later by MAL in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
- MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: MAL followed 4 hrs later by Ralt in Period 1, Ralt followed 4 hrs later by MAL in Period 2, Ralt alone in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
- Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: Ralt followed 4 hrs later by MAL in Period 1, Ralt alone in Period 2, MAL followed 4 hrs later by Ralt in Period 3, MAL followed 6 hrs later by Ralt in Period 4, Ralt followed 6 hrs later by MAL in Period 5
- Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: Ralt alone in Period 1, Ralt followed 4 hrs later by MAL in Period 2, MAL followed 4 hrs later by Ralt in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
- MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: MAL followed 4 hrs later by Ralt in Period 1, Ralt alone in Period 2, Ralt followed 4 hrs later by MAL in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
- Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt: Part 1 was comprised of Periods 1, 2 and 3; Period 3 was followed by a Pause of up to 37 days, before Part 2; Part 2 was comprised of Periods 4 and 5. Each period was separated by a washout of at least 2 days. Each Period had single oral dose treatments as follows: Ralt followed 4 hrs later by MAL in Period 1, MAL followed 4 hrs later by Ralt in Period 2, Ralt alone in Period 3, Ralt followed 6 hrs later by MAL in Period 4, MAL followed 6 hrs later by Ralt in Period 5
Period: Part 1 - Period 1
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 - Period 2
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 - Period 3
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 2 (One participant missed treatment during Period 3 only.) | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Pause (up to 37 Days)
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 3 (The participant who missed treatment in Period 3, resumed the study) | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2 - Period 4
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - Period 5
Arm/Group | Ralt-MAL4Ralt-Ralt4MAL-MAL6Ralt-Ralt6MAL | MAL4Ralt-Ralt4MAL-Ralt-MAL6Ralt-Ralt6MAL | Ralt4MAL-Ralt-MAL4Ralt-MAL6Ralt-Ralt6MAL | Ralt-Ralt4MAL-MAL4Ralt-Ralt6MAL-MAL6Ralt | MAL4Ralt-Ralt-Ralt4MAL-Ralt6MAL-MAL6Ralt | Ralt4MAL-MAL4Ralt-Ralt-Ralt6MAL-MAL6Ralt
Started | 3 | 3 | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All enrolled participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Raltegravir at 12 Hours (C 12 Hrs) in Part 1
Description: Blood was drawn 12 hours after dosing with raltegravir in order to determine the geometric mean plasma concentration.
Time Frame: 12 hours after dosing on Day 1 of each period
Population: The per-protocol population consisting of participants from Part 1 only, who complied with the study procedure and had available data from at least one treatment. One participant did not complete one period of Maalox-4 hour-Raltegravir treatment, resulting in an n = 17.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Groups:
- Raltegravir: 400 mg Raltegravir alone
- Maalox → 4 Hours → Raltegravir: 20 mL Maalox followed 4 hrs later by 400 mg Raltegravir
- Raltegravir → 4 Hours → Maalox: 400 mg Raltegravir followed 4 hrs later by 20 mL Maalox
Arm/Group | Raltegravir | Maalox → 4 Hours → Raltegravir | Raltegravir → 4 Hours → Maalox
Number analyzed (Participants) | 18 | 17 | 18
nM | 241.35 [177.31 to 328.52] | 96.29 [73.48 to 126.18] | 92.22 [72.31 to 117.60]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 4 Hours → Raltegravir; The hypothesis is that the true Raltegravir C 12 hrs geometric mean ratio (GMR) is not less than 0.4; Test type: Superiority or Other; p = 0.507, Hochberg step-up procedure; Geometric Mean Ratio (GMR) = 0.40, 90% CI 2-sided [0.31 to 0.52] — The Maalox followed by Raltegravir treatment group was the numerator, and the Raltegravir alone treatment group was the denominator
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 4 Hours → Maalox; The hypothesis is that the true Raltegravir C 12 hrs GMR is not less than 0.4; Test type: Superiority or Other; p = 0.624, Hochberg step-up procedure; GMR = 0.38, 90% CI 2-sided [0.30 to 0.49] — The Raltegravir followed by Maalox treatment group was the numerator, and the Raltegravir alone treatment group was the denominator

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC 0-12 Hrs) of Raltegravir in Part 1
Description: Blood was drawn at time 0, and at various intervals up to 12 hours after dosing with raltegravir in order to determine the geometric mean area under the curve plasma concentration versus time.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr.nM
Arm/Group | Raltegravir | Maalox → 4 Hours → Raltegravir | Raltegravir → 4 Hours → Maalox
Number analyzed (Participants) | 18 | 17 | 18
hr.nM | 17055.21 [11625.30 to 25021.30] | 13881.87 [9703.09 to 19860.30] | 11602.02 [7072.82 to 19031.55]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 4 Hours → Raltegravir; Test type: Superiority or Other; GMR = 0.81, 90% CI 2-sided [0.63 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 4 Hours → Maalox; Test type: Superiority or Other; GMR = 0.68, 90% CI 2-sided [0.50 to 0.92] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Maximum Plasma Concentration (C Max) of Raltegravir in Part 1
Description: Blood was drawn at time 0, and at various intervals up to 12 hours after dosing with raltegravir, in order to determine the geometric mean maximum plasma concentration.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir | Maalox → 4 Hours → Raltegravir | Raltegravir → 4 Hours → Maalox
Number analyzed (Participants) | 18 | 17 | 18
nM | 4723.00 [2837.48 to 7861.45] | 3690.96 [2321.28 to 5868.82] | 3324.84 [1829.19 to 6043.40]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 4 Hours → Raltegravir; Test type: Superiority or Other; GMR = 0.78, 90% CI 2-sided [0.55 to 1.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 4 Hours → Maalox; Test type: Superiority or Other; GMR = 0.70, 90% CI 2-sided [0.48 to 1.04] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Plasma Concentration of Raltegravir at 12 Hours (C 12 Hrs) in Part 2
Description: Blood was drawn 12 hours after dosing with raltegravir in order to determine the geometric mean plasma concentration.
Time Frame: 12 hours after dosing on Day 1 of each period
Population: The per-protocol population consisting of participants from the Raltegravir alone treatment group from Part 1, and the treatment groups from Part 2, who complied with the study procedure and had available data from at least one treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Groups:
- Maalox → 6 Hours → Raltegravir: 20 mL Maalox followed 6 hrs later by 400 mg Raltegravir
- Raltegravir → 6 Hours → Maalox: 400 mg Raltegravir followed 6 hrs later by 20 mL Maalox
Arm/Group | Raltegravir | Maalox → 6 Hours → Raltegravir | Raltegravir → 6 Hours → Maalox
Number analyzed (Participants) | 18 | 16 | 16
nM | 241.35 [178.78 to 325.83] | 121.52 [93.99 to 157.11] | 122.39 [101.28 to 147.90]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 6 Hours → Raltegravir; The hypothesis is that the true Raltegravir C 12 hrs GMR is not less than 0.4; Test type: Superiority or Other; GMR = 0.50, 90% CI 2-sided [0.39 to 0.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 6 Hours → Maalox; The hypothesis is that the true Raltegravir C 12 hrs GMR is not less than 0.4; Test type: Superiority or Other; GMR = 0.51, 90% CI 2-sided [0.40 to 0.64] — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC 0-12 Hrs) of Raltegravir in Part 2
Description: Blood was drawn at time 0, and at various intervals up to 12 hours after dosing with raltegravir, in order to determine the geometric mean area under the curve plasma concentration versus time.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1 of each period
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: hr.nM
Arm/Group | Raltegravir | Maalox → 6 Hours → Raltegravir | Raltegravir → 6 Hours → Maalox
Number analyzed (Participants) | 18 | 16 | 16
hr.nM | 17055.21 [11505.21 to 25282.47] | 14799.48 [10295.71 to 21273.38] | 15104.15 [10314.37 to 22118.22]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 6 Hours → Raltegravir; Test type: Superiority or Other; GMR = 0.87, 90% CI 2-sided [0.64 to 1.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 6 Hours → Maalox; Test type: Superiority or Other; GMR = 0.89, 90% CI 2-sided [0.64 to 1.22] — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Maximum Plasma Concentration (C Max) of Raltegravir in Part 2
Description: as for outcome 3
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1 of each period
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir | Maalox → 6 Hours → Raltegravir | Raltegravir → 6 Hours → Maalox
Number analyzed (Participants) | 18 | 16 | 16
nM | 4723.00 [2825.62 to 7894.45] | 4268.72 [2660.89 to 6848.07] | 4256.01 [2587.69 to 6999.93]
Statistical Analysis 1: Comparison: Raltegravir vs Maalox → 6 Hours → Raltegravir; Test type: Superiority or Other; GMR = 0.90, 90% CI 2-sided [0.58 to 1.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Raltegravir vs Raltegravir → 6 Hours → Maalox; Test type: Superiority or Other; GMR = 0.90, 90% CI 2-sided [0.58 to 1.41] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Up to 84 days
Description: Participants who received at least one dose of the investigational drug. Adverse events are reported not by the sequence of treatments, but rather by the treatment administered at the time of the adverse event.
Arm/Group | Raltegravir | Maalox → 4 Hours → Raltegravir | Raltegravir → 4 Hours → Maalox | Maalox → 6 Hours → Raltegravir | Raltegravir → 6 Hours → Maalox
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 1/17 | 1/18 | 2/16 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=18) | Maalox → 4 Hours → Raltegravir (N=17) | Raltegravir → 4 Hours → Maalox (N=18) | Maalox → 6 Hours → Raltegravir (N=16) | Raltegravir → 6 Hours → Maalox (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.